CLINICAL TRIAL: NCT01139957
Title: Prospective Study of Risk-Reducing Salpingo-Oophorectomy (RRSO) and Longitudinal CA-125 Screening Among Women at Increased Genetic Risk of Ovarian Cancer: Extended Follow-Up of Select GOG-0199 Study Participants
Brief Title: Incidence of Cancer in Women at Increased Genetic Risk of Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-8199; NCI-2011-02233 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000674216; GOG-8199 (Other: Gynecologic Oncology Group); GOG-8199 (Other: DCP); GOG-8199 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Breast Carcinoma; Fallopian Tube Carcinoma; Ovarian Neoplasm; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ancillary-correlative: Patients complete the Health Update Questionnaire annually for up to 5 years. The questionnaire focuses specifically on cancer risk, incidence, and mortality. Patients also receive ongoing communication (e.g., periodic newsletters, copies of study-related publications, etc.) to keep them informed regarding study-related research results, new research findings, new research opportunities for which patients may be eligible, and evolving clinical recommendations regarding hereditary breast/ovarian cancer.
  Interventions: Procedure: Evaluation of Cancer Risk Factors; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Study of High Risk Factors

INTERVENTIONS:
Procedure: Evaluation of Cancer Risk Factors — Ancillary studies
  Other Names: cancer risk factors evaluation
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Study of High Risk Factors — Ancillary studies

SUMMARY:
This clinical trial is studying the incidence of cancer in women at increased genetic risk of ovarian cancer. Gathering information about genetic factors in women with an increased risk of ovarian cancer over time may help doctors learn more about the disease and find better methods of treatment and on-going care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the prospective incidence of ovarian cancer, fallopian tube cancer, breast cancer, primary peritoneal cancer, and all cancer among women at increased risk of ovarian cancer, with a special emphasis on women who are known breast cancer susceptibility gene (BRCA)1/2 mutation carriers.

II. To develop precise point estimates of these cancer rates among women who have undergone risk-reducing salpingo-oophorectomy and women who have elected screening.

III. To compare the cancer rates between these two groups of women. IV. To better characterize the similarities and differences in cancer risk between BRCA mutation-positive families and BRCA mutation-negative/family history-positive families.

V. To develop preliminary estimates of overall and cancer-specific mortality, stratified by mutation status (BRCA1-positive, BRCA2-positive, BRCA1/2-negative).

OUTLINE: This is a multicenter study.

Patients complete the Health Update Questionnaire annually for up to 5 years. The questionnaire focuses specifically on cancer risk, incidence, and mortality. Patients also receive ongoing communication (e.g., periodic newsletters, copies of study-related publications, etc.) to keep them informed regarding study-related research results, new research findings, new research opportunities for which patients may be eligible, and evolving clinical recommendations regarding hereditary breast/ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled on GOG-0199

  * Completed the original 5-year follow-up period OR is off-study due to pregnancy or development of a new cancer
  * Completed the Off-Study form (Form Q0-0199 submitted via SEDES)
  * No patients who were off-study before the end of the initial 5-year follow-up period (found to be ineligible or consent withdrawal)

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the GOG-0199 protocol
Sampling Method: Probability Sample
Enrollment: 1916 (Estimated)
Dates: Start 2010-06-07 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Prospective incidence of ovarian cancer (including fallopian tube cancer), primary peritoneal cancer, breast cancer, and all cancer | Up to 5 years
Ovarian cancer mortality rates | Up to 5 years
  Cox proportional hazards models will be used to compare the incidence rates between the risk-reducing salpingo-oophorectomy (RRSO) and screening groups, adjusting for appropriate covariates. If necessary, modeling will be carried out in order to use non-proportional hazards models.
Breast cancer mortality rates | Up to 5 years
Quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Greene, Principal Investigator — Gynecologic Oncology Group
Locations (141):
- United States (141):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin